CLINICAL TRIAL: NCT05410717
Title: Phase I Trial to Evaluate Safety and Preliminary Efficacy of CLDN6/GPC3/Mesothelin/AXL-CAR-NK in Patients With CLDN6/GPC3/Mesothelin/AXL-positive Advanced Solid Tumors
Brief Title: CLDN6/GPC3/Mesothelin/AXL-CAR-NK Cell Therapy for Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZZCARNK-017
Record Dates: First submitted 2022-06-05; First posted 2022-06-08 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Stage IV Ovarian Cancer; Testis Cancer, Refractory; Endometrial Cancer Recurrent; CAR NK
Keywords: Solid tumor; Claudin6; CAR NK; GPC3; Mesothelin; AXL; Cannabidiol; Nicotinamide adenine dinucleotide; IL7; CCL19; PD1 antibody; PDL1 antibody; CTLA1 antibody
MeSH Terms: conditions — Ovarian Neoplasms; Testicular Neoplasms | interventions — claudin 6; Mesothelin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CAR-NK cell therapy group (Experimental): Appropriate patients who could benefit from the Claudin6, GPC3, Mesothelin, or AXL targeting CAR-NK cell therapy against solid cancers are chosen to be the CAR-NK cell therapy group.
  Interventions: Biological: Claudin6, GPC3, Mesothelin, or AXL targeting CAR-NK cells
- IL7/CCL19 secreting CAR-NK cell therapy group (Experimental): Appropriate patients who could benefit from the Claudin6, GPC3, Mesothelin, or AXL targeting CAR-NK cell therapy against solid cancers are chosen to be the IL7/CCL19 secreting CAR-NK cell therapy group.
  Interventions: Biological: Claudin6, GPC3, Mesothelin, or AXL targeting CAR-NK cells
- PD1/PDL1/CTLA4-scfv secreting CAR-NK cell therapy group (Experimental): Appropriate patients who could benefit from the Claudin6, GPC3, Mesothelin, or AXL targeting CAR-NK cell therapy against solid cancers are chosen to be the PD1/PDL1/CTLA4-scfv secreting CAR-NK cell therapy group.
  Interventions: Biological: Claudin6, GPC3, Mesothelin, or AXL targeting CAR-NK cells
- CAR-NK cell plus CBD therapy group (Experimental): Appropriate patients who could benefit from the Claudin6, GPC3, Mesothelin, or AXL targeting CAR-NK cell therapy against solid cancers are chosen to be the CAR-NK cell plus CBD therapy group.
  Interventions: Biological: Claudin6, GPC3, Mesothelin, or AXL targeting CAR-NK cells
- CAR-NK cell plus NAD therapy group (Experimental): Appropriate patients who could benefit from the Claudin6, GPC3, Mesothelin, or AXL targeting CAR-NK cell therapy against solid cancers are chosen to be the CAR-NK cell plus NAD therapy group.
  Interventions: Biological: Claudin6, GPC3, Mesothelin, or AXL targeting CAR-NK cells

INTERVENTIONS:
Biological: Claudin6, GPC3, Mesothelin, or AXL targeting CAR-NK cells — Engineering Claudin6, GPC3, Mesothelin, or AXL targeting CAR combined with/or without IL7/CCL19 and/or scfv against PD1/CTLA4/Lag3 secreting vector into NK cells, which are isolated from patients with advanced ovarian cancer or other cancers with expression of Claudin6, GPC3, Mesothelin, or AXL, and then transfusing them back the patients.
  In some cases, the CAR-NK cells will be combined with CBD or NAD to enhance the therapeutic efficacy.

SUMMARY:
This study is an open, exploratory clinical study to evaluate the safety and preliminary efficacy of Claudin6, GPC3, Mesothelin, or AXL targeting CAR-NK cells in patients with Claudin6, GPC3, Mesothelin, or AXL-positive advanced solid tumors (ovarian cancer and others)

DETAILED DESCRIPTION:
1. Choose appropriate advanced cancer patients with Claudin6, GPC3, Mesothelin, or AXL expression, with written consent for the study;
2. Perform PBMCs apheresis from the patient and isolate NK cells, transfect the NK cells with Claudin6, GPC3, Mesothelin, or AXL targeting CAR, amplify the number of transfected NK cells as needed, test the quality and killing activity of the Claudin6, GPC3, Mesothelin, or AXL-CAR-NK cells and then transplant back the patients via systemic or local infusions (via artery or intra-tumor), and follow up closely to collect related results as needed;
3. To enhance the killing capability, some CAR-NK cells are genetically engineered to express and secret IL7/CCL19 and/or SCFVs against PD1/CTLA4/Lag3; some CAR-NK cells are combined with Cannabidiol(CBD) or Nicotinamide adenine dinucleotide (NAD);
4. Evaluate the clinical results as needed.
5. Will also perform the similar clinical trial on different cancer types with Claudin6, GPC3, Mesothelin, or AXL expression.

ELIGIBILITY:
Inclusion Criteria:

1. patients with advanced ovarian cancer or other cancers with expression of claudin6.
2. Life expectancy >12 weeks
3. Adequate heart,lung,liver,kidney function
4. Available autologous transduced NK cells with greater than or equal to 20% expression of Claudin6, GPC3, Mesothelin, or AXL-CAR determined by flow-cytometry and killing of claudin6-positive targets greater than or equal to 20% in cytotoxicity assay
5. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent. -

Exclusion Criteria:

1. Had accepted gene therapy before;
2. Tumor size more than 25cm;
3. Severe virus infection such as HBV,HCV,HIV,et al
4. Known HIV positivity
5. History of liver/renal transplantation
6. Active infectious disease related to bacteria, virus,fungi,et al
7. Other severe diseases that the investigators consider not appropriate;
8. Pregnant or lactating women
9. Systemic steroid treatment (greater than or equal to 0.5 mg prednisone equivalent/kg/day)
10. Other conditions that the investigators consider not appropriate. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2036-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety by Common Terminology Criteria for Adverse Events (CTCAE) V5.0 | After CAR-NK cells infusion, up to 52 weeks.
  The type, frequency, severity, and duration of adverse events as a result of Claudin6, GPC3, Mesothelin, or AXL- CAR-NK cells infusion will be summarized.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | After CAR-NK cells infusion, up to 52 weeks.
  Per Response Evaluation Criteria in Solid Tumours (RECIST 1.1) assessed by MRI or CT. ORR defined as the proportion of patients in whom a complete response (CR) or partial response (PR) is observed as best overall response, prior to progression or further anti-cancer therapy.
Disease control rate (DCR) | up to 52 weeks.
  Disease control rate (DCR) defined as the proportion of patients in whom a CR or PR or stable disease (SD) (per RECIST 1.1, SD assessed at least 6 weeks after the first dose) is observed as best overall response.
Duration of response (DOR) | up to 36 months
  Duration of response (DOR) defined as the time from first objective response (CR or PR per RECIST 1.1) to first occurrence of objective tumor progression (Progressive disease (PD) per RECIST 1.1/recurrence) or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD, PHD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No